CLINICAL TRIAL: NCT00004998
Title: A Phase II, Open-Label Study of AG1549 in Combination With Other Antiretroviral Agents in Treatment-Naive HIV-Infected Patients
Brief Title: Safety and Effectiveness of a New Anti-HIV Drug (AG1549) in Combination With Other Anti-HIV Drugs in HIV-Infected Patients
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 286B; AG1549-503
Record Dates: First submitted 2000-03-21; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Nelfinavir; Combivir
MeSH Terms: conditions — HIV Infections | interventions — lamivudine, zidovudine drug combination; capravirine; Nelfinavir

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Capravirine
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to see if two different doses of AG1549 plus other anti-HIV drugs are safe and effective in HIV-infected patients who are not taking anti-HIV drugs.

DETAILED DESCRIPTION:
[Note: As of 2/28/2001, due to toxicity studies and concerns for safety, sites were notified that they need to discontinue patients from the capravirine/placebo arms and continue patients with their background therapies or switch patients to new therapies, as deemed appropriate by the investigators.] Patients are randomized to receive one of two doses of AG1549 plus Viracept (nelfinavir) plus Combivir (zidovudine/lamivudine). Patients remain on their assigned therapy for 48 weeks, with a follow-up visit at 28 to 35 days after the last dose of study medication. Blood samples are taken regularly to quantify HIV-1 RNA, CD4 and CD8 counts, peripheral blood mononuclear cells (PBMC), AG1549, Viracept, and M8 plasma concentrations. Physical exams, safety assessments, and other tests are also done throughout the study. On Day 8 and at the end of Week 48, pharmacokinetic samples are collected at 0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, and 12.0 hours postdose. At the end of Weeks 4, 8, 16, 24, and 36, pharmacokinetic samples are taken prior to dosing and between 2 to 4 hours post-dose.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible if they:

* Are HIV-positive.
* Are at least 18 years old.
* Have a CD4 cell count of more than 50 cells/mm3.
* Have an HIV level of more than 5000 copies/ml.

Exclusion Criteria

Patients will not be eligible if they:

* Have ever taken any of the following anti-HIV drugs: nonnucleoside reverse transcriptase inhibitors (NNRTIs), AG1549, Viracept, zidovudine, lamivudine, or Combivir. Other anti-HIV drugs are allowed only if taken for no more than 30 days with the last dose taken more than 6 months prior to study entry.
* Have taken an experimental drug within 28 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Clin Research of West Florida, Clearwater, Florida
  - Community Health Care, Fort Lauderdale, Florida
  - South Shore Hosp, Miami, Florida
  - Infectious Diseases Associates, Sarasota, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Catholic Med Ctr, Jamaica, New York
  - Liberty Medical, New York, New York
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
- Immunity Care and Research Inc, Santo Domingo, Dominican Republic